CLINICAL TRIAL: NCT01133691
Title: Examination of Gastric Emptying With Magnetic Resonance Imaging and Ultrasonography
Brief Title: Examination of Gastric Emptying in Children
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2009-0147
Record Dates: First submitted 2010-05-11; First posted 2010-05-31 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Gastric Emptying
Keywords: gastric emptying; children; gastric fluid volume; preoperative fasting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy children aged 6 - 12 years
  Interventions: Dietary Supplement: clear fluid, light breakfast

INTERVENTIONS:
Dietary Supplement: clear fluid, light breakfast — clear fluid 7 ml/kg, breakfast consisting of yoghurt, muesli, mild

SUMMARY:
* Background: Fasting is mandatory for safety of anesthesia in elective surgery and imaging but gives rise to discomfort, hunger and thirst especially in children. Internationally accepted fasting times are often prolonged because of organisational delay in operating theatre.
* Hypothesis: Clear fluids can be ingested until an imaginary anesthesia induction time without enlarging the residual gastric contents compared to overnight fast. There is no difference between residual gastric contents after 4 hours of fasting after a light meal compare to 6 hours in healthy children.
* Examination of gastric volume using magnetic resonance imaging after overnight fasting and subsequent scans after either clear fluid intake or intake of a standard breakfast are performed in children aged 6 - 12 years. Time course after fluid intake is followed with scans every half hour for 2 hours. In the breakfast group 4 versus 6 hours fasting time will be simulated, e. g. intake of clear fluid is allowed for 2 versus 4 hours after the meal. Volume of gastric contents will be compared with a standardized ultrasonographic view of the stomach.

ELIGIBILITY:
Inclusion Criteria:

* age 6 - 12 years
* ASA I or II

Exclusion Criteria:

* gastrointestinal pathology
* claustrophobia
* implants like pacemaker, ventriculoperitoneal shunt etc
* symptomatic or relevant cardiac, renal or metabolic disease

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy children aged 6 - 12 years old
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Gastric emptying time | 6 hours
  Time after food/fluid ingestion when gastric volume after overnight fast is achieved, as measured by volumetry of magnetic resonance scans

SECONDARY OUTCOMES:
gastric volume after fasting | 6 hours
gastric antral area | 6 hours
visual analog scale of thirst/hunger | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Achim J Schmitz, MD, Principal Investigator — Children's University Hospital Zurich, Anesthesiology
Locations (1):
- University Children's Hospital, Anesthesiology, Zurich, Canton of Zurich, Switzerland